CLINICAL TRIAL: NCT00800150
Title: Phase I Study of Escalating Doses of Radiation Therapy Using Helical Tomotherapy in Combination With Fludarabine (FLU) and Melphalan (MEL) as a Preparative Regimen for Allogeneic Hematopoietic Stem Cell (HSC) Transplantation in Patients With Advanced and Hematological Malignancies Who Are Not Eligible for Fully Myeloablative Regimen
Brief Title: Total Marrow and Total Lymph Node Irradiation, Fludarabine, and Melphalan Followed By Donor Stem Cell Transplant in Treating Patients With Advanced Hematological Cancer That Has Not Responded to Treatment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol objective could not be met. A new study with amended eligibility criteria will be developed.
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 08076; P30CA033572 (NIH); CHNMC-08076; CDR0000626148 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-11-27; First posted 2008-12-01 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; splenic marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III mycosis fungoides/Sezary syndrome; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV mycosis fungoides/Sezary syndrome; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; primary myelofibrosis; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; cutaneous B-cell non-Hodgkin lymphoma; Waldenstrom macroglobulinemia
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Congenital Abnormalities; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Intraocular Lymphoma; Primary Myelofibrosis; Waldenstrom Macroglobulinemia | interventions — fludarabine phosphate; Melphalan; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fludarabine phosphate
Drug: melphalan
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation
Radiation: intensity-modulated radiation therapy
Radiation: tomotherapy
Radiation: total marrow irradiation
Radiation: total nodal irradiation

SUMMARY:
RATIONALE: Giving total marrow and total lymph node irradiation together with low doses of chemotherapy before a donor stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect).

PURPOSE: This phase I trial is studying the side effects and best dose of total marrow and total lymph node irradiation when given together with fludarabine and melphalan followed by donor stem cell transplant in treating patients with advanced hematological cancer that has not responded to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of intensity-modulated total marrow and lymph node irradiation (TMLI) using helical tomotherapy in combination with a reduced-intensity preparative regimen comprising fludarabine phosphate and melphalan in patients undergoing allogeneic hematopoietic stem cell transplantation for advanced, relapsed or refractory hematological malignancies.
* To describe the toxicities of escalating doses of TMLI in these patients.

Secondary

* To describe the frequency of clinical response in patients treated with this regimen.
* To describe the frequency of primary and secondary engraftment failure in patients treated with this regimen.
* To describe the time to neutrophil and platelet engraftment in patients treated with this regimen.
* To describe the incidence of acute and chronic graft-versus-host disease in patients treated with this regimen.
* To describe the overall survival of patients treated with this regimen.
* To describe the progression-free survival of patients treated with this regimen.

OUTLINE: This is a dose-escalation study of intensity-modulated total marrow and lymph node irradiation (TMLI).

* Intensity-modulated radiation therapy: Patients undergo TMLI to skeletal bone/marrow, major lymph node chains, spleen, and liver using helical tomotherapy twice daily on days -6 to -3.
* Reduced-intensity preparative regimen: Patients receive fludarabine phosphate IV on days -6 to -2 and melphalan IV on day -1.
* Hematopoietic stem cell transplantation (HSCT): Patients undergo allogeneic HSCT on day 0.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histopathologically confirmed diagnosis of 1 of the following:

  * Acute myeloid leukemia (AML)
  * Myelodysplastic syndromes

    * Intermediate- or high-risk disease
  * Myelofibrosis
  * Granulocytic sarcoma (chloroma)

    * With or without bone marrow involvement
  * Mixed lineage leukemia

    * Induction therapy must have been directed predominantly against AML
  * Acute lymphoblastic leukemia
  * Non-Hodgkin lymphoma
  * Multiple myeloma
* Relapsed or refractory disease with M3 marrow (marrow blasts > 25%), meeting 1 of the following criteria:

  * Persistent disease after an induction attempt
  * Persistent initial disease after two induction attempts
  * Relapse after one re-induction attempt (second relapse)
  * Persistent disease after first relapse and initial re-induction attempt
* Not eligible for myeloablative allogeneic hematopoietic stem cell transplantation due to age (> 50 years), organ insufficiency, or significant comorbidity

  * Patients 16-50 years of age must meet ≥ 1 of the following criteria:

    * Ejection fraction 50-60% by MUGA scan and/or echocardiogram
    * DLCO 50-75% of predicted
    * Creatinine clearance or GFR 60-80 mL/min
    * Serum bilirubin ≤ 2.0 mg/dL
    * SGOT and SGPT 1.5-5 times upper limit of normal
    * No other medical and/or psychosocial problem that, in the opinion of the primary physician or principal investigator, would place the patient at unacceptable risk from study regimen
* No Fanconi anemia
* HLA-identical sibling OR matched unrelated donor available

PATIENT CHARACTERISTICS:

* Zubrod or Karnofsky performance status 70-100%
* Negative pregnancy test
* Able to lie supine in a full body cast for 30 minutes
* No HIV infection
* No evidence of active hepatitis B or C infection
* No evidence of cirrhosis
* No uncontrolled viral, bacterial, or fungal infection within the past 4 weeks
* No radiographic changes indicating pulmonary disease (e.g., pulmonary nodules, infiltrates, or pleural effusion) unless cleared by pulmonary biopsy that shows no evidence of active pulmonary disease
* No major medical or psychiatric disorder that would seriously compromise patient tolerance of study regimen

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiation therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of intensity-modulated total marrow and lymph node irradiation using helical tomotherapy
Toxicity

SECONDARY OUTCOMES:
Frequency of clinical response
Frequency of primary and secondary engraftment failure
Time to neutrophil and platelet engraftment
Incidence of acute and chronic graft-versus-host disease
Overall survival
Progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Rosenthal, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States